CLINICAL TRIAL: NCT00230503
Title: Dose-Ranging Study of Pradefovir in Patients With Compensated Hepatitis B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RNA200103-201
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis B, Chronic; Hepatitis B Virus; Pradefovir Mesylate; Adefovir Dipivoxyl
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — pradefovir

INTERVENTIONS:
Drug: pradefovir mesylate
Drug: adefovir dipivoxyl

SUMMARY:
* Compare the safety of four oral doses of pradefovir after 48 weeks of treatment
* Select the dose of pradefovir for Phase 3 studies

DETAILED DESCRIPTION:
* Compare the safety of four oral doses of pradefovir after 48 weeks of treatment
* Compare the antiviral activity of four oral doses of pradefovir to adefovir and dipivoxyl after 48 weeks of treatment
* Select the dose of pradefovir for Phase 3 studies
* Determine the pharacokinetic profiles of four oral doses of pradefovir

ELIGIBILITY:
Inclusion Criteria:

* Compensated chronic HBV Infection
* No prior treatment with adefovir dipivoxil
* No interferon or lamivudine treatment for three months prior to enrollment
* HBeAg positive or negative
* HBV DNA viral load greater than 500,000 copies per mL
* ALT between 1.2 and 10 times ULN

Exclusion Criteria:

* Positive HIV, HCV, and/or HDV serology
* History of renal tubular necrosis
* Serum creatinine greater than 2.0 mg/dl
* History of organ transplant or use of immunosuppresive drugs
* Pregnant or breast-feeding females

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220
Dates: Start 2004-06; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
- Safety: Clinical examinations of laboratory tests
- Efficacy: Change in viral load over time

SECONDARY OUTCOMES:
- Efficacy: Proportion of patients with undetectable viral load

CONTACTS AND LOCATIONS:
Overall Officials: Ralph T. Doyle, Study Director — Bausch Health Americas, Inc.

REFERENCES:
- [Derived] Gao Y, Kong F, Song X, Shang J, Yao L, Xia J, Peng Y, Liu W, Gong H, Mu M, Cui H, Han T, Chen W, Wu X, Yang Y, Yan X, Jin Z, Wang P, Zhu Q, Chen L, Zhao C, Zhang D, Jin W, Wang D, Wen X, Liu C, Jia J, Mao Q, Ding Y, Jin X, Zhang Z, Mao Q, Li G, Niu J. Pradefovir Treatment in Patients With Chronic Hepatitis B: Week 24 Results From a Multicenter, Double-Blind, Randomized, Noninferiority, Phase 2 Trial. Clin Infect Dis. 2022 Jun 10;74(11):1925-1932. doi: 10.1093/cid/ciab763. PMID 34487151